CLINICAL TRIAL: NCT03442660
Title: Psychometric Validation Study of the Spasticity Quality of Life 6-Dimensions (SQOL-6D) in Upper-limb Spasticity
Brief Title: Validation of the Spasticity Related Quality of Life Questionnaire
Acronym: SQOL-6D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: F-FR-52120-232
Record Dates: First submitted 2017-12-15; First posted 2018-02-22 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Spasticity, Muscle
MeSH Terms: conditions — Muscle Spasticity | interventions — Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Data collection (Other): An electronic data capture (EDC) system will be used to collect data in electronic format. Data will be collected at the enrolment visit, at the follow-up visit (8 weeks +/-2 weeks) and 1 to 4 days after the follow-up visit.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Subjects will be treated in accordance with usual medical practice during their participation in this study. No additional diagnostic or treatment procedures will be required. Subjects will be asked to complete electronic (or on paper when it's not possible to use electronic version) questionnaires.

SUMMARY:
The purpose of the study is to describe the psychometric properties (validity, reliability and responsiveness) of the SQOL-6D instrument in the context of routine clinical treatment of upper limb spasticity.

DETAILED DESCRIPTION:
The study qualifies as interventional not because of the use of an investigational product, but because the imposed specific data collection procedures include multiple questionnaire assessments and one on-site visit not necessarily part of routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Currently resident in the UK
* Subjects with a diagnosis of ULS
* Receiving a treatment at the enrolment visit, as part of their routine clinical management, aiming at reducing spasticity
* Sufficient grasp of English and cognitive ability to be able to understand the SQOL-6D questions, give informed consent and complete the protocol requirements as judged by the investigator

Exclusion Criteria:

* The subject has already been included in the study
* The subject, in the opinion of the investigator, would be unable to understand the questionnaire or to comply with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Validation of SQOL-6D in upper limb spasticity | Change from baseline (day 1) to 8 weeks +/-2 weeks (follow up visit)
  Validity - Reliability - Responsiveness

SECONDARY OUTCOMES:
EQ-5D-5L (EuroQoL 5 Dimensions, 5 Levels) | Day 1 and then 8 weeks +/-2
  A summary index score will be calculated from responses given to the 5 domain items, measuring overall health on a scale 0 to 1 using United Kingdom (UK) value sets.
Neurological Impairment Scale adapted for ULS (ULS-NIS) | Day 1
  Records functional impairment on a four-point scale (rated 0-3) across seven domains, including: motor impairment in the affected upper limb, sensation affected in the affected upper limb, communication, cognitive function, cortical function, emotional/behaviour and mobility of joints, as measured by soft tissue shortening (an assessment used for the evaluation of the deterioration in range of movement due to spasticity by percentage loss of range).
Modified Ashworth Scale (MAS) | Day 1 and then 8 weeks +/-2
  Six-point scale (with available scores of 0, 1, 1+, 2, 3 and 4) evaluates muscle tone by reporting changes in this during muscle flexion or extension, depending on the (resistance in) joint mobility being assessed (shoulder, elbow, wrist or finger).
Gaseous (Goal Attainment Scaling Evaluation of Outcome for Upper-Limb Spasticity) | Day 1 and then 8 weeks +/-2
  Goal attainment will be recorded on a five point numerical scale (range -2 to +2) and goal scores combined to give an aggregated T score.
ArmA (Arm Activity Measure) Scores | Day 1 and then 8 weeks +/-2
  ArmA is a patient-reported outcomes questionnaire recording the difficulty in caring for, and completing tasks and activities with the affected arm. The ArmA contains a total of 29 items in four subscales. Difficulty for each item is assessed on a five-point scale (range 0 to 4).
Global assessment of benefit | 8 weeks +/-2
  The Global Assessment of Benefit scale will be completed by the subject. Responses options will be: Much worse (-2)/Worse (-1)/Same (0)/Some benefit (+1)/Great benefit (+2).

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (8):
- United Kingdom (8):
  - Hull and East Yorkshire NHS Trust, Castle Hill Hospital, Cottingham
  - Mid Yorkshire Hospitals NHS Trust, Dewsbury Hospital, Dewsbury
  - London North West NHS Healthcare Trust - Regional Hyper-acute Rehabilitation Unit, Harrow
  - University Hospitals of Leicester NHS Trust, Neurology Department, Leicester General Hospital, Leicester
  - Northumberland Tyne and Wear NHS trust, Walkergate Park Neuro-Rehabilitation, Newcastle
  - Staffordshire and Stoke-on-Trent Partnership NHS Trust, North Staffordshire Rehabilitation Centre, Haywood Hospital, Stoke-on-Trent
  - City Hospitals Sunderland NHS Foundation Trust Research and Innovation Education Centre, Sunderland
  - South Warwickshire NHS Foundation Trust, Central England Rehabilitation Unit Leamington Spa Hospital, Warwick

REFERENCES:
- [Derived] Turner-Stokes L, Fheodoroff K, Jacinto J, Lambert J, De La Loge C, Calvi-Gries F, Whalen J, Lysandropoulos A, Maisonobe P, Ashford S. The spasticity-related quality of life 6-dimensions instrument in upper-limb spasticity: Part I Development and responsiveness. J Rehabil Med. 2022 Jan 3;54:jrm00244. doi: 10.2340/jrm.v53.690. PMID 34726763